CLINICAL TRIAL: NCT01216423
Title: Is There a Link Between Venous Thromboembolism and Stroke in Patient With Patent Foramen Ovale ? Research for Stroke in Hospitalized Patients With Pulmonary Embolism.
Brief Title: Pulmonary Embolism and Stroke in Patient With Patent Foramen Ovale
Acronym: EPIC-FOP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC-FOP
Record Dates: First submitted 2010-09-29; First posted 2010-10-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Recent Stroke; Pulmonary Embolism; Patent Foramen Ovale
Keywords: Patent Foramen Ovale; Pulmonary embolism; Stroke
MeSH Terms: conditions — Pulmonary Embolism; Foramen Ovale, Patent; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Incidence of recent stroke in patients with PFO
- Incidence of recent stroke in patients without PFO

SUMMARY:
The cause of ischemic stroke remains frequently unknown. In patients with patent foramen ovale (PFO), the link between PFO and Stroke is unclear. The investigators hypothesize that the main mechanism is paradoxical embolism and decided to look for clinically apparent and silent cerebral embolism in patients with a recent pulmonary embolism.

DETAILED DESCRIPTION:
Inclusion criteria :

* age > 18 years old
* confirmed pulmonary embolism
* informed consent
* social ensured

Exclusion criteria :

* pregnancy
* age < 18 years old
* protected major person (in sense of public health)
* consent refused
* MRI contraindications

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* confirmed pulmonary embolism
* informed consent
* social ensured

Exclusion Criteria:

* pregnancy
* age < 18 years old
* protected major person (in sense of public health)
* consent refused
* MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of hospitalized patients with pulmonary embolism
Sampling Method: Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2009-11; Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of recent ischemic stroke in patients hospitalized for a recent pulmonary embolism with comparison in two groups with and without PFO | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle LE MOIGNE, MD, Principal Investigator — University Hospital, Brest
Locations (4):
- France (4):
  - Army Hospital, Brest, France
  - CHU Dijon de Bocage, Dijon, France
  - Centre Hospitalier de Cornouaille, Quimper, France
  - Brest University Hospital, Brest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Moigne E, Timsit S, Ben Salem D, Didier R, Jobic Y, Paleiron N, Le Mao R, Joseph T, Hoffmann C, Dion A, Rousset J, Le Gal G, Lacut K, Leroyer C, Mottier D, Couturaud F. Patent Foramen Ovale and Ischemic Stroke in Patients With Pulmonary Embolism: A Prospective Cohort Study. Ann Intern Med. 2019 Jun 4;170(11):756-763. doi: 10.7326/M18-3485. Epub 2019 May 7. PMID 31060047